CLINICAL TRIAL: NCT04531826
Title: The Use of Five-strand Hamstring Autograft to Increase the Graft Size in Anterior Cruciate Ligament Reconstruction - a Prospective Randomized Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital Authority, Hong Kong (Other Government)
Responsible Party: Principal Investigator, Keith Hay-Man Wan, Associate Consultant, Hospital Authority, Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HAREC1
Record Dates: First submitted 2020-08-26; First posted 2020-08-31 (Actual); Last update posted 2020-08-31 (Actual); Status verified 2020-08

CONDITIONS: Anterior Cruciate Ligament Injuries
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): Five-strand hamstring autograft group
  Interventions: Other: 5-strand hamstring graft preparation
- Group B (Placebo Comparator): Quadripled hamstring autograft group
  Interventions: Other: 5-strand hamstring graft preparation

INTERVENTIONS:
Other: 5-strand hamstring graft preparation — Five-strand hamstring graft preparation

SUMMARY:
Anterior cruciate ligament (ACL) reconstruction is one of most commonly performed orthopaedic surgeries. Several options for graft choice are available and autologous single bundle hamstring graft is most commonly used. Variability exists among patients in terms of hamstring size, and therefore the graft diameter. Recently there has been an increasing amount of literature correlating the hamstring graft diameter with the graft failure rate [1-4]. They concluded that graft exceeding 8mm in diameter is associated with a significant lower risk of graft failure. There has been study showing that Asian patients were indeed 'different' from the Caucasians. Ho et al published his findings on Singaporean patients showing that the median graft diameters for female and male patients were 7mm and 8mm respectively [5]. A retrospective review our patients undergoing ACL reconstruction in our department over the past 10 years has shown that the mean graft diameter was 7.8mm (range, 5.5-10mm).

The conventional way of four-strand hamstring autograft is done by doubling both the semitendinosus and gracilis tendons to provide a quadrupled graft. Several techniques have been described to increase the size of the hamstring graft. One of those is the -strand hamstring graft, in which the longer semitendinosus tendon is tripled with the shorter gracilis tendon doubled to produce a 5-strand configuration. We hypothesized that the 5-strand hamstring graft would provide a graft of significantly larger diameter than the conventional quadrupled autograft.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-50
* Symptoms and physical examinations consistent with ACL deficiency and magnetic resonance imaging indicating ACL injury

Exclusion Criteria:

* Previous surgeries in the operated knee
* Revision ACL reconstruction
* Contralateral ACL injury
* Concomitant posterior cruciate ligament / collateral ligament surgeries in the operated knee

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 62 (Estimated)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Mean graft diameter | Intra-operative

SECONDARY OUTCOMES:
Adverse event | Post-operative 3 months, 6 months, 9 months, 12 months, 18 months and 2 years.
  intra-operative complications, infections, venous thromboembolism
ACL failure | Post-operative 3 months, 6 months, 9 months, 12 months, 18 months and 2 years.
  Graft failure / re-rupture, ACL revision, contralateral ACL injury
Clinical measures of knee function and structure | Post-operative 3 months, 6 months, 9 months, 12 months, 18 months and 2 years.
  strength testing, hoop test, range of motion, knee osteoarthritis.

IPD SHARING:
Plan to Share IPD: Undecided